CLINICAL TRIAL: NCT00431262
Title: Antabuse in Severe Alcoholism: an Open Controlled Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Psykiatrisk Center Gentofte (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT no. 2006-004921-27
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2007-03-05 (Estimated); Status verified 2007-03

CONDITIONS: Alcoholism
Keywords: alcoholism; antabuse; disulfiram; abstinence; cognitive behavioural therapy
MeSH Terms: conditions — Alcoholism | interventions — Disulfiram

INTERVENTIONS:
Drug: antabuse (disulfiram)

SUMMARY:
Newly detoxified alcoholics (N=60) are randomised to either antabuse (disulfiram) treatment or the control group for a total of 6 months.All patients will receive cognitive behavioural treatment in groups. The hypothesis to be tested is that more of the patients who receive antabuse (disulfiram) will be alcohol free during the 6 months treatment period compared to the control group. The trial is open.

ELIGIBILITY:
Inclusion Criteria:

* Alcoholism
* Living in the departments catchment area

Exclusion Criteria:

* Pregnancy
* Schizophrenia
* Bipolar disorder
* Other substance abuse
* Dementia
* Anorexia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2007-02; Study Completion 2009-06

PRIMARY OUTCOMES:
The number of patients in each group who have not been drinking alcohol after 6 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Ulrichsen, MD, ph.d., Principal Investigator — Psykiatrisk Center Gentofte
Locations (1):
- Psykiatrisk Center Gentofte, Hellerup, Denmark